CLINICAL TRIAL: NCT02364258
Title: Pharmacokinetics of Rosuvastatin and Atorvastatin in Pediatric Dyslipidemia Patients: Clinical Impact of Genetic Variation in Statin Disposition
Brief Title: Pharmacokinetics of Rosuvastatin and Atorvastatin in Pediatric Dyslipidemia Patients
Acronym: SD2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jon Wagner, Pediatric Cardiologist/Clinical Pharmacology, Children's Mercy Hospital and Clinics, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13020063
Record Dates: First submitted 2015-02-03; First posted 2015-02-18 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 10mg tablet (ages 8-21 years); 1 time dose given per oral at the start of the study day.
  Interventions: Drug: Rosuvastatin
- Atorvastatin (Experimental): Atorvastatin 10mg tablet (ages 8-21 years); 1 time dose given per oral at the start of the study day.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 10mg tablet (ages 8-21 years); 1 time dose given per oral at the start of the study day.
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Atorvastatin — Atorvastatin 10mg tablet (ages 8-21 years); 1 time dose given per oral at the start of the study day.
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
This will be a single center, open label, randomized, cross-over study in patients with dyslipidemia comparing the pharmacokinetics of rosuvastatin and atorvastatin in patients with greater than or equal to one variant allele in the SLCO1B1 gene (-11187 and/or c.521) to patients with the wild-type/wild-type genotype.

The studies goal is to establish the role of genetic variation and development in key transporters on the dose-exposure relationship of two commonly used statin drugs in children. This study is the first step in a series of investigations aimed to determining the mechanisms behind variations in physiologic response, clinical efficacy and significant adverse effect risk that surround the statin drugs in children and adolescents.

DETAILED DESCRIPTION:
Trial Design

Investigational Agents:

Rosuvastatin 10mg tablet (ages 8-21 years); oral dosing Atorvastatin 10mg tablet (ages 8-21 years); oral dosing Commercial supplies of rosuvastatin and atorvastatin that are FDA approved for use in pediatric dyslipidemia will be used. Rosuvastatin and atorvastatin from the same source and lot will be used for all subjects.

Dose Rationale:

The doses designated above are chosen according to previous pediatric data13,14, and are consistent with current labeling for rosuvastatin and atorvastatin in children greater than 10 years of age. The rosuvastatin and atorvastatin doses will be off label for participants 8-10 years of age, but consistent with current practice. Data from this study are not intended to be used to change the drug labeling, and thus a new IND is not required. Although fixed doses within a pre-specified age range will be used, dose data will be analyzed corrected for weight (mg/kg) based on the patient's weight at time of dosing.

Risk/Benefits:

All eligible subjects with a LDL >130mg/dl (95% percentile) meet current clinical criteria for statin therapy. The risks associated with participation in this single-dose pharmacokinetic study are expected to be minimal given the known adverse event profile for the study articles and also, the limited exposure. The most common mild adverse effects of statins are headache, myalgia, and gastrointestinal symptoms (abdominal pain, dyspepsia, diarrhea, constipation). However, in children these adverse effects occur with the same frequency as placebo7,10,25. Rare adverse effects include elevation of hepatic transaminases and myopathy, but these are generally observed with chronic treatment. Furthermore, no cases of hepatic failure with statins have been reported to date10. There is also a small risk associated with placement of the intravenous (IV) catheter that will be used to draw serial blood samples for pharmacokinetic analysis and screening/safety labs. Finally, there is the risk of loss of confidentiality for the participating subjects. Methods to protect PHI and data handling are specifically outlined in the CMH CPR protocol Sections 4 & 5 (CMH IRB# 12040220). All of the above risks associated with this non-therapeutic clinical trial are minimal.

There is no direct benefit to participating subjects, although there may be benefit for children in the future, as it is expected that the information to be gained from the study can be generalized to the larger population of pediatric patients who may require statin treatment. The purpose of the study is to determine how genetic variation impacts rosuvastatin and atorvastatin plasma concentrations following recommended doses of the drug in a patient population that has not previously been studied. Thus, with this knowledge, future protocols could subsequently be developed to effectively "personalize" dosing for pediatric subjects with the aforementioned SNPs who are taking rosuvastatin and atorvastatin, thereby improving efficacy and safety for the individual patient.

Study Design/Type:

This will be a single center, open-label, randomized, crossover pilot study in patients with dyslipidemia comparing the pharmacokinetics of rosuvastatin and atorvastatin in patients with greater than or equal to one variant allele in the SLCO1B1 gene (-11187 and/or c.521) to patients with the wild-type/wild-type genotype. The results of genetic testing will not be disclosed to the subjects.

Population Sample:

The CMH Cardiology Pharmacogenomics Repository (CPR) (CMH IRB# 12040220) database will be accessed to determine subjects meeting inclusion/exclusion criteria. The study population from the aforementioned IRB proposal has already agreed to be contacted for future studies. Once the target population and an equal set of age, sex-, race- and Tanner Stage-matched controls are identified, the patients will be invited to participate.

Subject Recruitment:

Once a target population and an equal set of age-, sex- and Tanner Stage-matched controls are identified from the CPR, prospective participants will be informed about the study. Initial contact will occur by way of a prepared telephone script (Appendix 2&3). Those that agree to participate will be scheduled for a visit to the Pediatric Clinical Research Unit (PCRU) for a screening visit. At this visit, the study will be explained to the patient/patient's family, permission/assent/consent (Appendix 4&5) will be obtained, a physical examination (including Tanner staging), and screening laboratory testing will be performed. Participants for whom permission/assent/consent has been obtained and inclusion criteria are met, will be scheduled to come back to the PCRU for the first study drug day. If the participant is currently on a statin, they will not be scheduled to come back for at least 6 days for Study Drug Day #1 (washout period). This visit will need to be conducted following a minimum of 6 days and up to 14 days for these participants. If the participant is not currently on a statin then they can be scheduled anytime after their screening visit is complete. The visit will consist of a physical examination, lab tests, placement of an indwelling venous cannula for serial blood draws as outlined below and administration of a single oral dose of rosuvastatin or atorvastatin. The total amount of blood drawn (screening labs and PK samples) for the trial will be 60.6 ml, which is well within the guidelines placed at CMH ORI for children > 25 kg. This study will require an overnight stay in the PCRU in order to obtain all necessary plasma levels. Following a minimum of 6 days and up to 14 days after the study day #1 (washout period), the participating subject will be brought back to the PCRU for another single dose pharmacokinetic study involving the second drug with the same procedure and sampling scheme as conducted in study day #1.

ELIGIBILITY:
Inclusion Criteria:

1. Children 8-21 years of age
2. LDL cholesterol >130mg/dl (>95% percentile)
3. Successfully genotyped for SLCO1B1
4. Willing to sign the assent/permission/consent form

Exclusion Criteria:

1. Underlying structural heart disease including congenital heart disease or acquired heart disease.
2. History or laboratory evidence of an underlying intestinal, metabolic, autoimmune, or renal disease that could alter the disposition of rosuvastatin or atorvastatin.
3. Underlying pathology of the gastrointestinal tract or recent surgery which would be expected to alter the rate and/or extent of drug absorption
4. Evidence of previous hypersensitivity to statin medications
5. Unwillingness or inability to have screening labs drawn
6. Refusal to participate in the study
7. Unwillingness or inability to participate in an overnight fast
8. Subjects taking drugs with interactions with statins (CYP3A4 inducers/inhibitors, OATP1B1 inducers/inhibitors) (Appendix 1)
9. Inability to swallow a tablet drug
10. For females, a positive urine beta-human chorionic gonadotropin pregnancy test result
11. Evidence of hepatic abnormality as determined by values > 3 times the age-specific upper limit of normal for AST, ALT, total and conjugated bilirubin, serum albumin, Alkaline Phosphatase, and GGT.
12. Abnormal red blood cell morphology and/or a hemoglobin less than 9 gm/dl
13. Diarrhea in the last 24 hours

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Evaluate effect of genotype (SLCO1BI) on Cmax rosuvastatin | 2 years
Evaluate effect of genotype (SLCO1B1) on AUC rosuvastatin | 2 years
Evaluate effect of genotype (SLCO1BI) on Cmax atorvastatin | 2 years
Evaluate effect of genotype (SLCO1B1) on AUC atorvastatin | 2 years

SECONDARY OUTCOMES:
Evaluate the effect of age on Cmax of rosuvastatin | 2 years
Evaluate the effect of gender on Cmax of rosuvastatin | 2 years
Evaluate the effect of race on Cmax of rosuvastatin | 2 years
Evaluate the effect of sexual maturity on Cmax of rosuvastatin | 2 years
Evaluate the effect of age on Cmax of atorvastatin | 2 years
Evaluate the effect of age on AUC of atorvastatin | 2 years
Evaluate the effect of gender on AUC of atorvastatin | 2 years
Evaluate the effect of race on AUC of atorvastatin | 2 years
Evaluate the effect of sexual maturity on AUC of atorvastatin | 2 years
Evaluate the effect of age on AUC of rosuvastatin | 2 years
Evaluate the effect of gender on AUC of rosuvastatin | 2 years
Evaluate the effect of race on AUC of rosuvastatin | 2 years
Evaluate the effect of sexual maturity on AUC of rosuvastatin | 2 years
Evaluate the effect of age on Ka of atorvastatin | 2 years
Evaluate the effect of gender on Ka of atorvastatin | 2 years
Evaluate the effect of race on Ka of atorvastatin | 2 years
Evaluate the effect of sexual maturity on Ka of atorvastatin | 2 years
Evaluate the effect of age on Ka of rosuvastatin | 2 years
Evaluate the effect of gender on Ka of rosuvastatin | 2 years
Evaluate the effect of race on Ka of rosuvastatin | 2 years
Evaluate the effect of sexual maturity on Ka of rosuvastatin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jon B Wagner, DO, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States